CLINICAL TRIAL: NCT06576440
Title: The Effects of Ghrelin Administration on Motivation and Resting Energy Expenditure
Brief Title: Effects of Ghrelin Administration on Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: TUE008_ADMIN
Record Dates: First submitted 2024-08-21; First posted 2024-08-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder
Keywords: energy homeostasis; motivation; ghrelin; anhedonia; mood
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia | interventions — Ghrelin; acyl-ghrelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Major depressive disorder (Experimental): Patients with major depressive disorder will receive a subcutaneous injection of ghrelin (experimental) on one day and saline (placebo) on another day (order randomised; double-blind cross-over design).
  Interventions: Drug: Ghrelin; Drug: Saline
- Healthy control participants (Experimental): Healthy control participants will receive a subcutaneous injection of ghrelin (experimental) on one day and saline (placebo) on another day (order randomised; double-blind cross-over design).
  Interventions: Drug: Ghrelin; Drug: Saline

INTERVENTIONS:
Drug: Ghrelin — Participants in this arm will receive a subcutaneous injection of acyl-ghrelin as the active condition.
  Other Names: Acyl-ghrelin
Drug: Saline — Participants in this arm will receive a subcutaneous injection of saline as placebo control condition.
  Other Names: Placebo

SUMMARY:
Everyday humans are confronted with a plethora of rewards competing for their attention. Nevertheless, to obtain a goal or reward, humans often need to invest effort. When humans are confronted with the challenge to integrate costs of action such as the effort of walking to one's favorite lunch place with its anticipated benefits (i.e., eating one's favorite meal), accumulating evidence suggest that humans might "go with the gut". Ghrelin is a stomach-derived hormone and the only known circulating peptide that stimulates appetite. At the same time, patients with major depressive disorder report deficits in motivated behavior which are oftentimes accompanied by changes in appetite and weight. Based on a wealth of accruing evidence from animal studies, the investigators suggest that the gut acts as an important arbitrator in effort allocation by signaling the energy level of the body. Within this physiological framework, ghrelin is thought to signal a short-term energy deficit to increase reward responsivity and willingness to work for reward as compensatory (allostatic) means. Here, the investigators propose to conduct a follow-up study (to NCT05318924) with subcutaneous administration of ghrelin vs. saline in patients with major depressive disorder and healthy control participants. During each visit, participants will receive a subcutaneous administration of either ghrelin or saline and perform an effort allocation task where they have to exert physical effort to obtain food and monetary rewards. The investigators hypothesize that ghrelin will increase the motivation to exert effort for rewards. The goal of this follow-up study is to test that the motivational effects of ghrelin are similar in patients with depression and healthy control participants. Furthermore, participants resting energy expenditure will be estimated before and after the administration. In line with a role of ghrelin as an energy deficit signal, the investigators expect ghrelin to decrease energy expenditure. During each visit, participants will answer questions about their current mood and physiological state. The investigators hypothesize that ghrelin increases mood state and hunger while decreasing satiety.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in the behavioral study arm of NCT05120336

Exclusion Criteria:

* participation in the neuroimaging part of NCT05120336
* breastfeeding
* pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Ghrelin-induced changes in motivation | 15-50 minutes after subcutaneous administration (ghrelin vs. saline)
  Frequency of button presses on a XBox controller to obtain rewards after ghrelin administration vs. saline administration
Ghrelin-induced changes in Resting Energy Expenditure | Pre injection versus 50-65 minutes after injection (compared to saline)
  Changes in energy expenditure after a ghrelin administration (vs. saline) as measured with indirect Calorimetry.
Ghrelin-induced changes in mood | Pre injection timepoints (mean over 40 minutes and 5 minutes before) versus post injection timepoints (mean over 15, 50 and 65 minutes after injection) (compared to saline)
  Changes operationalized via visual analogue ratings (0-100) of the sum score of positive and negative affect schedule mood items after ghrelin administration vs. saline administration. Measures are taken ~40 minutes and 5 minutes prior to injection, as well as 15, 50, and 65 minutes after injection.
Ghrelin-induced changes in hunger and satiety from baseline | Pre injection timepoints (mean over 40 minutes and 5 minutes before) versus post injection timepoints (mean over 15, 50 and 65 minutes after injection) (compared to saline)
  Change in visual analogue scale (0-100) measures of subjective hunger and satiety after ghrelin administration vs. saline administration. Measures are taken ~40 minutes and 5 minutes prior to injection, as well as 15, 50, and 65 minutes after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Nils B Kroemer, PhD, Principal Investigator — University of Tübingen, Faculty of Medicine, Department of Psychiatry & Psychotherapy
Locations (1):
- Department of Psychiatry & Psychotherapy, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, behavioral data will be shared after aggregation at the trial or participant level.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access